CLINICAL TRIAL: NCT00277810
Title: A 6-Month, Randomized, Double-Blind, Placebo-Controlled, Multicenter, Safety, Tolerability, and Efficacy Study of 3 Doses of Lecozotan (SRA-333) SR in Outpatients With Mild to Moderate Alzheimer's Disease Treated With a Cholinesterase Inhibitor
Brief Title: Study Evaluating the Safety, Tolerability, and Efficacy of Lecozotan SR in Outpatients With Alzheimer's Disease
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 3098B1-203, 3098B1-204
Record Dates: First submitted 2006-01-12; First posted 2006-01-16 (Estimated); Last update posted 2020-07-07 (Actual); Status verified 2020-07

CONDITIONS: Alzheimer Disease
Keywords: Alzheimer's Disease; Cholinesterase Inhibitors; Outpatients
MeSH Terms: conditions — Alzheimer Disease | interventions — lecozotan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- A (Experimental)
  Interventions: Drug: lecozotan SR (SRA-333)
- B (Experimental)
  Interventions: Drug: lecozotan SR (SRA-333)
- C (Experimental)
  Interventions: Drug: lecozotan SR (SRA-333)

INTERVENTIONS:
Drug: lecozotan SR (SRA-333) — one of 3 doses of lecozotan sr dose for 6 months as an extension to a 6 month study with patients required to be on a cholinesterase inhibitor 2, 5, or 10 mg of lecozotan sr

SUMMARY:
The purpose of the study is to determine the safety, tolerability, and efficacy of 3 doses of lecozotan in combination with a cholinesterase inhibitor in patients with mild to moderate Alzheimer's disease (AD).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of probable Alzheimer's disease
* Current use of cholinesterase inhibitor
* Able to give signed and dated informed consent and lives with appropriate caregiver at home or in community dwelling with caregiver accompanying patient to all visits and visiting patient at least daily for duration of the study

Exclusion Criteria:

* Significant neurological disease other than AD
* Diagnosis of major depression
* History of stroke or other heart disease

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2006-03; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
All events and physical and neurological function and score change from baseline to 24 weeks in ratings for cognitive and global function scales | 6 mo extension study: week 24

SECONDARY OUTCOMES:
Score change from baseline to 24 weeks on functional and behavioral scales | week 24

CONTACTS AND LOCATIONS:
Locations (77):
- United States (33):
  - Phoenix, Arizona
  - Tucson, Arizona
  - Costa Mesa, California
  - Fresno, California
  - La Jolla, California
  - Orange, California
  - Delray Beach, Florida
  - Fort Lauderdale, Florida
  - Fort Myers, Florida
  - Hallandale, Florida
  - Hialeah, Florida
  - Jacksonville, Florida
  - Miami, Florida
  - Miami Beach, Florida
  - Orlando, Florida
  - Sarasota, Florida
  - South Miami, Florida
  - Tampa, Florida
  - West Palm Beach, Florida
  - St Louis, Missouri
  - Long Branch, New Jersey
  - Manchester Twp., New Jersey
  - Albany, New York
  - Cedarhurst, New York
  - Staten Island, New York
  - Winston-Salem, North Carolina
  - Columbus, Ohio
  - Tulsa, Oklahoma
  - Philadelphia, Pennsylvania
  - East Providence, Rhode Island
  - Memphis, Tennessee
  - Houston, Texas
  - Bennington, Vermont
- Argentina (9):
  - Av. Belgrano
  - Buenos Aires
  - Calle Adolfo Alsina
  - Cervino
  - Gascon
  - Larrea
  - Nueva York
  - Pilar
  - Puerto Galván
- Australia (5):
  - Adelaide
  - East Gosford
  - Hornsby
  - Randwick
  - Victoria
- Canada (5):
  - Edmonton, Alberta
  - Medicine Hat, Alberta
  - Moncton, New Brunswick
  - Ottawa, Ontario
  - Montreal, Quebec
- Finland (3):
  - Helsinki
  - Joensuu
  - Kuopio
- France (4):
  - Bordeaux
  - Montpellier
  - Nice
  - Toulouse
- Roma, Italy
- Poland (6):
  - Gdansk - Wrzeszcz
  - Krakow
  - Lodz
  - Lublin
  - Sopot
  - Szczecin
- South Africa (4):
  - Bloemfontein
  - Cape Town
  - Johannesburg
  - Somerset West
- Spain (2):
  - Barcelona
  - Madrid
- United Kingdom (5):
  - Belfast
  - Glasgow
  - Sheffield
  - Southampton
  - Swindon